CLINICAL TRIAL: NCT04316832
Title: A Randomized-Controlled Trial: the Effectiveness of a Single-session of Mindfulness Based Cognitive Training on CVC and Core Symptoms in Children and Adolescents With ADHD
Brief Title: Mindfulness Based Cognitive Training in Children and Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Andeea Robe, Principal investigator, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Phd study ARobe
Record Dates: First submitted 2020-03-11; First posted 2020-03-20 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: ADHD
Keywords: ADHD; mindfulness based cognitive training; cardiac vagal control; children and adolescents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This will be a two-arm, randomized controlled trial exploring whether a single-session of MBIs could improve task-related scores of attention, mood and CVC in children and adolescents with ADHD/ADD referred to a Romanian Child and Adolescent Psychiatric Unit. Outcomes assessment will be conducted at baseline, immediately after the session of training (T1) and 4 weeks after the intervention (T2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation will be implemented using a random numbers generator, https://www.random.org/lists/. The allocation ratio will be 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/treatment (Experimental): The mindfulness based cognitive training will be delivered in one session and will include short mindfulness exercises.
  Interventions: Behavioral: Mindfulness based cognitive training
- No intervention (Placebo Comparator): Control exercise, participants will listen to the first chapter of the audiobook The Hobbit, JRR Tolkien.
  Interventions: Other: Control exercise

INTERVENTIONS:
Behavioral: Mindfulness based cognitive training — The mindfulness based cognitive training will include three short mindfulness exercises: a) a breathing exercise, b) a body scan exercise, and c) a mindfulness attention exercise.
  Arms: Intervention/treatment
Other: Control exercise — Participants will listen to the first chapter of the audiobook The Hobbit, JRR Tolkien.
  Arms: No intervention

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is one of the most common neurodevelopmental disorders, with a pooled worldwide prevalence of 7.2% among children. Although medication and behavioral therapy, have been shown to be effective for reducing core symptoms, about 30% of patients with ADHD would not achieve the treatment response and symptomatic remission. Additionally, some children can experience sides effects related to medication. Therefore, other psychological approaches such as Mindfulness based interventions (MBIs) have been designed for the management of ADHD.

Recent research showed that ADHD is associated with autonomic nervous system dysregulation, characterized by reduced vagally mediated-HRV, in response to a task demand. HRV is an accurate, non-invasive, cost-effective quantitative biomarker of autonomic nervous system (ANS) activity. There is evidence that MBIs could significantly reduce ADHD core symptoms and may enhance HRV through increased parasympathetic modulation. No studies have jointly examined the differential effect of MBIs on ADHD core symptoms, task related-HRV and mood.

The aim of this study is to assess the effectiveness of a single-session of mindfulness based cognitive training on CVC, core symptoms and mood in children and adolescents with ADHD, aged 6 y-17y, referred to an outpatient Romanian Child and Adolescent Psychiatric Unit by mental health professionals, teachers and/or parents.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is one of the most common neurodevelopmental disorders, with a pooled worldwide prevalence of 7.2% among children. Children/adolescents with ADHD face significant disease burden; they experience poorer academic achievement and attainment, higher rates of risky sexual practices and early unwanted pregnancies, increase risk of substance use and relationship difficulties. Although medication and behavioral therapy, particularly given by parents and with active child and teacher involvement, have been shown to be effective for reducing core symptoms, about 30% of patients with ADHD would not achieve the treatment response and symptomatic remission. Additionally, some children can experience sides effects related to medication such as sleep problem or weight loss. Therefore, other psychological approaches such as Mindfulness based interventions (MBIs), have been designed for the management of ADHD.

Heart rate variability (HRV) represents the oscillation in time between successive heartbeats, and it can be evaluated by time- and frequency-domain measures. Recent research showed that ADHD is associated with autonomic nervous system dysregulation, characterized by reduced vagally mediated-HRV, in response to a task demand. HRV is an accurate, non-invasive, cost-effective quantitative biomarker of autonomic nervous system (ANS) activity.

Over the years, research has cumulated for supporting the use of mindfulness for various clinical health conditions. There is evidence that MBIs could significantly reduce ADHD core symptoms and may enhance HRV through increased parasympathetic modulation.

Although emerging research has shown that mindfulness has led to improvements in the core symptoms of ADHD, most of the research in this area involves extensive multi week trainings; there is limited research evaluating brief mindfulness programs in the context. Therefore, the aim of this study is to assess the effectiveness of a single-session of mindfulness based cognitive training on CVC, core symptoms and mood in children and adolescents with ADHD, aged 6 y-17y.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of ADHD
* Able to verbally communicate and write in Romanian.
* Normal intellectual ability.
* Not taking any medication/No change in ADHD specific medication(dose/type) or psychological intervention within 3 months of trial onset.

Exclusion Criteria:

* Comorbidities of Conduct Disorder, ODD, OCD
* Other chronic diseases
* Previous participation in mindfulness-based training

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Reaction time (RT) to correct responses during a computerized Continuous performance tests (CPTs) | Change from baseline RT (time 0) at immediately after the intervention (time 1) and after additional 4 weeks after the intervention (time 2) .
  A non-x CPT task in wich the subjects must press the space bar for any letter but X. The RT measures the amount of time between the presentation of the stimulus and the client's response.
% Omission errors (OR) during a computerized Continuous performance tests (CPTs) | Change from baseline OR (time 0) at immediately after the intervention (time 1) and after additional 4 weeks after the intervention (time 2) .
  A non-x CPT task in wich the subjects must press the space bar for any letter but X. The OR indicates the number of times the target was presented, but the client did not respond/click the mouse.
% Commission errors (CR) during a computerized Continuous performance tests (CPTs) | Change from baseline CR (time 0) at immediately after the intervention (time 1) and after additional 4 weeks after the intervention (time 2) .
  A non-x CPT task in wich the subjects must press the space bar for any letter but X. The score of CR indicates the number of times the client responded but no target was presented.

SECONDARY OUTCOMES:
Vagally mediated heart rate variability (HRV)= Cardiac Vagal Control (CVC) | Change from baseline CVC (time 0) at immediately after the intervention (time 1) and after additional 4 weeks (time 2)
  The oscillation in time between successive heartbeats.
Mood | Change from baseline mood (time 0) at immediately after the intervention (time 1) and after additional 4 weeks (time 2)
  Mood will be evaluated through a 4 basic emotions, using a Visual Analogue Scale (VAS) (e.g., To what extent are you experiencing anxiety, sadness, anger or worry at this moment?'). A 10 cm (100 mm) horizontal line with verbal descriptors at each side of the line to express the extremes of the feeling (e.g., 'not at all' versus 'very much') will be used.

OTHER OUTCOMES:
The empirically based syndromes scales of the Child Behavioral Checklist (CBCL): Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Social Problems,Thought Problems, Attention Problems, Rule Breaking Behavior, Aggressive Behavior | Changes in time from baseline (time 0) at 4 weeks after the intervention '(time 2).
  Child Behavioral Checklist for Ages 6-18, (Achenbach & Rescorla, 2004) is The Child Behavior Checklist (CBCL) is a checklist parents complete to detect emotional and behavioural problems in children and adolescents. It consists of 113 questions, scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often).
Inattention (IA) subscale raw score and Hyperactivity- Impulsivity (HI) subscale raw score | Changes in time IA and HI subscale from baseline (time 0) at 4 weeks after the intervention (time 2)
  ADHD Rating Scale-IV: Parent Version; is a 18-questions questionnaire in which the parents rate the the frequency of a specific behavior related to innatention or hyperactivity-impulsivity using one of the following "always or very often", "often", "somewhat", or "rarely or never".

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Robe, Principal Investigator — UBB; Anca Dobrean, Study Director — UBB
Locations (1):
- S.C. Rega Med SRL, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beauchaine TP, Thayer JF. Heart rate variability as a transdiagnostic biomarker of psychopathology. Int J Psychophysiol. 2015 Nov;98(2 Pt 2):338-350. doi: 10.1016/j.ijpsycho.2015.08.004. Epub 2015 Aug 11. PMID 26272488
- [Background] Catala-Lopez F, Hutton B, Nunez-Beltran A, Page MJ, Ridao M, Macias Saint-Gerons D, Catala MA, Tabares-Seisdedos R, Moher D. The pharmacological and non-pharmacological treatment of attention deficit hyperactivity disorder in children and adolescents: A systematic review with network meta-analyses of randomised trials. PLoS One. 2017 Jul 12;12(7):e0180355. doi: 10.1371/journal.pone.0180355. eCollection 2017. PMID 28700715
- [Background] DuPaul, G. J., Power, T. J., Anastopoulos, A. D., & Reid, R. (1998). ADHD Rating Scale-IV: Checklists, norms, and clinical interpretation. Guilford Press.
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Graham J, Coghill D. Adverse effects of pharmacotherapies for attention-deficit hyperactivity disorder: epidemiology, prevention and management. CNS Drugs. 2008;22(3):213-37. doi: 10.2165/00023210-200822030-00003. PMID 18278977
- [Background] Hall CL, Valentine AZ, Groom MJ, Walker GM, Sayal K, Daley D, Hollis C. The clinical utility of the continuous performance test and objective measures of activity for diagnosing and monitoring ADHD in children: a systematic review. Eur Child Adolesc Psychiatry. 2016 Jul;25(7):677-99. doi: 10.1007/s00787-015-0798-x. Epub 2015 Nov 30. PMID 26620873
- [Background] Howarth, A., Smith, J. G., Perkins-Porras, L., & Ussher, M. (2019). Effects of Brief Mindfulness-Based Interventions on Health-Related Outcomes: A Systematic Review. 10, 1957-1958. https://doi.org/10.1007/s12671-019-01163-1
- [Background] Kramer RS, Weger UW, Sharma D. The effect of mindfulness meditation on time perception. Conscious Cogn. 2013 Sep;22(3):846-52. doi: 10.1016/j.concog.2013.05.008. Epub 2013 Jun 15. PMID 23778017
- [Background] Robe A, Dobrean A, Cristea IA, Pasarelu CR, Predescu E. Attention-deficit/hyperactivity disorder and task-related heart rate variability: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2019 Apr;99:11-22. doi: 10.1016/j.neubiorev.2019.01.022. Epub 2019 Jan 24. PMID 30685483
- [Background] Zou L, Sasaki JE, Wei GX, Huang T, Yeung AS, Neto OB, Chen KW, Hui SS. Effects of Mind(-)Body Exercises (Tai Chi/Yoga) on Heart Rate Variability Parameters and Perceived Stress: A Systematic Review with Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2018 Oct 31;7(11):404. doi: 10.3390/jcm7110404. PMID 30384420
- [Background] Xue J, Zhang Y, Huang Y. A meta-analytic investigation of the impact of mindfulness-based interventions on ADHD symptoms. Medicine (Baltimore). 2019 Jun;98(23):e15957. doi: 10.1097/MD.0000000000015957. PMID 31169722
- [Background] Thomas R, Sanders S, Doust J, Beller E, Glasziou P. Prevalence of attention-deficit/hyperactivity disorder: a systematic review and meta-analysis. Pediatrics. 2015 Apr;135(4):e994-1001. doi: 10.1542/peds.2014-3482. Epub 2015 Mar 2. PMID 25733754
- [Background] Shim SH, Yoon HJ, Bak J, Hahn SW, Kim YK. Clinical and neurobiological factors in the management of treatment refractory attention-deficit hyperactivity disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Oct 3;70:237-44. doi: 10.1016/j.pnpbp.2016.04.007. Epub 2016 Apr 19. PMID 27103462
- [Result] Achenbach, T. M., & Rescorla, L. A. (2004). The Achenbach System of Empirically Based Assessment (ASEBA) for Ages 1.5 to 18 Years. In The use of psychological testing for treatment planning and outcomes assessment: Instruments for children and adolescents, Volume 2, 3rd ed. (pp. 179-213). Lawrence Erlbaum Associates Publishers.
- [Derived] Robe A, Dobrean A. The effectiveness of a single session of mindfulness-based cognitive training on cardiac vagal control and core symptoms in children and adolescents with attention-deficit/hyperactivity disorder (ADHD): a preliminary randomized controlled trial. Eur Child Adolesc Psychiatry. 2023 Oct;32(10):1863-1872. doi: 10.1007/s00787-022-02005-7. Epub 2022 May 24. PMID 35608666